CLINICAL TRIAL: NCT06552403
Title: Effect of a Modified 5:2 Intermittent Fasting Diet on Population With Overweight or Obesity in China: A Self-controlled Clinical Trial
Brief Title: Effect of a Modified 5:2 Intermittent Fasting Diet on Population With Overweight or Obesity in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Provincial Tongde Hospital (Other)
Responsible Party: Principal Investigator, Xiaoli Wang, Principal Investigator, Zhejiang Provincial Tongde Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5:2 intermittent fasting diet
Record Dates: First submitted 2024-07-31; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified 5:2 IF diet (Experimental): The modified 5:2 IF diet involves 2 nonconsecutive fasting days (25%-30% of the total required daily energy intake based on ideal body weight) and 5 days of habitual intake (limited total energy intake according to ideal body weight) per week, as well as a 4-week run-in period and a minimum of 6,000 steps of physical activity per day.
  Interventions: Dietary Supplement: A modified 5:2 intermittent fasting diet

INTERVENTIONS:
Dietary Supplement: A modified 5:2 intermittent fasting diet — The modified 5:2 IF diet involves 2 nonconsecutive fasting days (25%-30% of the total required daily energy intake based on ideal body weight) and 5 days of habitual intake (limited total energy intake according to ideal body weight) per week, as well as a 4-week run-in period and a minimum of 6,000 steps of physical activity per day.

SUMMARY:
This study aimed to investigate the effects of the modified 5:2 IF dietary intervention on the Chinese population with overweight or obesity based on a self-controlled clinical trial.

DETAILED DESCRIPTION:
There are fewer studies on the influence of dietary interventions on the Chinese populations with obesity, and the degree of obesity, body fat distribution, dietary pattern and structure, and metabolic status of populations with obesity are different between the Chinese and European populations. The effects of a 5:2 IF dietary intervention on the Chinese population with overweight or obesity are unclear. Therefore, this study aimed to investigate the effects of the modified 5:2 IF dietary intervention on the Chinese population with overweight or obesity based on a self-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. participants aged 18 to 60 years
2. participants with a body mass index (BMI) ≥ 24 kg/m2
3. participants engaged in light physical labor and their weight was relatively stable.

Exclusion Criteria:

1. participants taking any medication with an effect on body weight in the three months prior to enrollment;
2. participants with liver or kidney dysfunction (liver enzymes ≥ 2 times normal; blood creatinine > the upper limit of normal);
3. participants with a history of cardiovascular disease (e.g., coronary heart disease, stroke);
4. participants with malignant tumors;
5. women during pregnancy or breastfeeding;
6. participants deemed unsuitable by the investigator to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
body measurements | 24 weeks after intervention
  weight, BMI, and waistline
glycolipid metabolism indicators | 24 weeks after intervention
  fasting plasma glucose (FPG), fasting plasma insulin (FPI), fasting C-peptide (FCP), triglycerides (TG), total cholesterol (TC), low density lipoprotein-cholesterol (LDL-C), high density lipoprotein-cholesterol (HDL-C), and uric acid.
adipokines | 24 weeks after intervention
  leptin and lipocalin
inflammatory factors before the modified 5:2 IF diet intervention and after 24 weeks of intervention | 24 weeks after intervention
  high sensitivity C-reactive protein (hsCRP), interleukin 6 (IL-6), and tumor necrosis factor-alpha (TNF-α)

SECONDARY OUTCOMES:
Change in metabolic components | 24 weeks after intervention
  Participants' metabolic components were analyzed by serum metabolomics analysis. The ultra-high performance liquid chromatography combined with quadrupole time-of-flight mass spectrometry (UPLC-QTOF-MS) (Agilent 1290, Agilent Technologies, Inc., USA) was applied to identify metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Wang, Principal Investigator — Zhejiang Provincial Tongde Hospital
Locations (1):
- Xiaoli Wang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No